CLINICAL TRIAL: NCT00095316
Title: A Randomized, Double-Masked Trial of Caspofungin Versus Placebo as Prophylaxis of Invasive Candidiasis in High-Risk Adults in the Critical Care Setting
Brief Title: Caspofungin Study for Fungal Infections in Adults in Critical Care Settings
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 02-042; BAMSG 2-01
Record Dates: First submitted 2004-11-02; First posted 2004-11-03 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2006-06

CONDITIONS: Candidiasis
Keywords: candidiasis, caspofungin, fungal infection, prophylaxis
MeSH Terms: conditions — Candidiasis; Mycoses | interventions — Caspofungin

ARMS (2):
- Placebo (Placebo Comparator): Subjects receive placebo intravenously daily for 28 days
  Interventions: Other: Placebo
- Caspofungin (Experimental): Subjects receive 50mg/day caspofungin intravenously (IV) for 28 days
  Interventions: Drug: Caspofungin

INTERVENTIONS:
Drug: Caspofungin — Caspofungin is an antifungal agent of the echinocandin class of glucan synthase inhibitor. Subjects receive Caspofungin acetate 50mg/day IV for 28 days.
  Arms: Caspofungin
Other: Placebo — Normal saline equivalent to that used to deliver the caspofungin given intravenously as a single daily dose infused over approximately 1 hour for 28 days
  Arms: Placebo

SUMMARY:
Adults admitted to intensive care units are at risk for a variety of complications. One of the most frequent complications is the development of new infections. Infections due to a fungus called Candida are of particular concern. This study will test the possibility that caspofungin, a new therapy for fungal infections, may reduce the rate of Candida infections in subjects at risk.

DETAILED DESCRIPTION:
A Randomized, Double-Masked Trial of Caspofungin (50 mg/day) Versus Placebo as Prophylaxis of Invasive Candidiasis in HighRisk Adults in the Critical Care Setting for up to 28 days with observation of primary outcome through 7 days after study therapy. The primary objective of this study is to evaluate the efficacy of caspofungin as prophylaxis for invasive candidiasis in high-risk ICU patients as opposed to those receiving placebo whereas the secondary objectives are as follows: To evaluate the utility of surrogate markers for the diagnosis of invasive candidiasis, to assess the effect of colonization as a risk factor in developing the disease, evaluate the safety of prophylactic caspofungin in subjects who discontinue the study due to drug-related adverse events versus subjects with 1 or more drug-related adverse events and to evaluate the all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

Non-pregnant subjects >/= 18 years of age; admission to the ICU during the preceding 3 days (minimum of 2 days in ICU) and expected to stay in the ICU a minimum of 2 additional days; subjects must have at least 1 of the following: received at least one other dose of any systemic antibiotic on any one of the ICU days before study entry and continue to receive antibiotics at the time of enrollment, and/or presence of a central venous catheter at the time of enrollment and for one additional day during the current ICU stay, and at least 2 of the following: use of total parenteral nutrition on any of Days 1-4 of ICU stay; any type of dialysis on any of Days 1-4 of ICU stay; any in-patient surgery done under general anesthesia or epidural block in the 7 days prior to or on ICU admission*; pancreatitis (documented by computed tomography (CT) scan or lipase >1,000 u/L) in the 7 days prior to or on ICU admission; more than 1 dose of systemic steroids (prednisone equivalent dose >/=20 mg per dose) in the 7 days prior to or on ICU admission; and/or use of more than 1 dose of other systemic immunosuppressive agents (such as azathioprine, tacrolimus, sirolimus, mycophenolate, monoclonal antibodies, and tumor necrosis factor [TNF] immunomodulators) in the 7 days prior to or on ICU admission.

* Excludes placement of vascular catheters.

Exclusion Criteria:

Subjects with an allergy or intolerance to caspofungin or other echinocandin analog; absolute neutrophil count <500/mm3 at entry or likely to develop such a count during therapy; diagnosis of HIV, aplastic anemia, or chronic granulomatous disease; moderate or severe hepatic insufficiency as defined by a Child Pugh score of 7 or greater or cirrhosis due to any cause; pregnancy or breastfeeding; subjects unlikely to survive more than 2 days; subjects who have received systemic antifungal therapy within 7 days prior to study entry; subjects with documented active, proven, or probable invasive fungal infection within 7 days prior to study entry; subjects previously enrolled into this trial; subjects currently receiving another investigational agent or who have received an investigational agent within the 7 days prior to study entry; subjects in the ICU 5 or more days prior to enrollment into this study .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2004-10; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - University of Alabama Hospital - Infectious Diseases, Birmingham, Alabama
  - University of Southern California - Infectious Diseases, Los Angeles, California
  - Harbor UCLA Medical Center - Medicine - Infectious Diseases, Torrance, California
  - University of Colorado Hospital - Denver, Denver, Colorado
  - MedStar Washington Hospital Center - Infectious Diseases, Washington D.C., District of Columbia
  - Jackson Memorial Hospital, Miami, Florida
  - Emory University School of Medicine - Infectious Diseases, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago College of Medicine - Infectious Diseases, Chicago, Illinois
  - The University of Chicago - Medicine - Infectious Diseases & Global Health, Chicago, Illinois
  - Loyola University - Emergency Facility, Maywood, Illinois
  - Infectious Disease of Indiana, PSC, Indianapolis, Indiana
  - University of Kentucky - UK Albert B Chandler Hospital, Lexington, Kentucky
  - Overton Brooks VA Medical Center, Shreveport, Louisiana
  - Mark Hatfield Clinical Research Center, Bethesda, Maryland
  - Tufts Medical Center - Infectious Diseases Clinic, Boston, Massachusetts
  - University of Michigan - VA Ann Arbor Health Care Systems, Ann Arbor, Michigan
  - Harper University Hospital, Detroit, Michigan
  - Henry Ford Health System - Henry Ford Hospital, Detroit, Michigan
  - University of Mississippi - Infectious Diseases, Jackson, Mississippi
  - Cooper University Hospital - Infectious Diseases, Camden, New Jersey
  - Duke University Medical Center - Duke Clinical Research Institute, Durham, North Carolina
  - Memorial Hermann Hospital, Houston, Texas
  - University of Texas Health Science Center at San Antonio - Infectious Diseases, San Antonio, Texas
  - University of Virginia Primary Health Center - Infectious Diseases and International Health, Charlottesville, Virginia
  - University of Wisconsin Hospital and Clinics - Clinical Science Center - Nephrology, Madison, Wisconsin